CLINICAL TRIAL: NCT01126554
Title: ICG- Liver Test Versus New Biomarkers as Prognostic Markers in Critically Ill
Brief Title: ICG- Liver Test Versus New Biomarkers as Prognostic Markers in Critically Ill Patients
Acronym: Greenpep
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Brahms AG (Industry)
Responsible Party: Sponsor
Other Study IDs: CIM_MB 002; CIM_02 (Other: KEK)
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Critically Ill
Keywords: Prognostic value
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Critically ill patients

SUMMARY:
Comparison of ICG liver testing with copeptin and SAPS II score as prognostic markers in critically ill patients.

DETAILED DESCRIPTION:
Comparison of different marker for length of stay in the ICU in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the ICU

Exclusion Criteria:

* Not able to understand German

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill patients of a 10 bed ICU unit
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
prolonged length of stay in the ICU (pLOS) more than 3 days | 3 days
  see above

CONTACTS AND LOCATIONS:
Overall Officials: Markus Béchir, MD, Principal Investigator — CIM
Locations (1):
- Surgical ICU, University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Zoller B, Spanaus K, Gerster R, Fasshauer M, Stehberger PA, Klinzing S, Vergopoulos A, von Eckardstein A, Bechir M. ICG-liver test versus new biomarkers as prognostic markers for prolonged length of stay in critically ill patients - a prospective study of accuracy for prediction of length of stay in the ICU. Ann Intensive Care. 2014 Jul 8;4:19. doi: 10.1186/s13613-014-0019-7. eCollection 2014. PMID 25045579